CLINICAL TRIAL: NCT06119984
Title: A Community-based Intervention to Address Social Norms Associated With Intimate Partner Violence in Rural Southwest, Nigeria
Brief Title: Community-based Intervention to Prevent Intimate Partner Violence in Rural Southwest, Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Funmilola OlaOlorun (Other)
Collaborators: University of Ibadan (Other)
Responsible Party: Sponsor-Investigator, Funmilola OlaOlorun, Senior Lecturer, University of Ibadan
Organization: University of Ibadan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SNIP Project
Record Dates: First submitted 2023-10-07; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Violence; Domestic Violence; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community mobilization (Experimental): a six-month community mobilization intervention that consisted of advocacy to stakeholders, community workshops and small group discussions in intervention communities
  Interventions: Behavioral: Community mobilization
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Community mobilization — The intervention focused on creating awareness, challenging social norms, and promoting actions against violence. To achieve these, the following activities were undertaken: introductory meetings, selection and training of model couples, structured workshops and small group meetings.
  Arms: Community mobilization

SUMMARY:
Background:

Intimate partner violence is arguably the most prevalent, persistent and pernicious type of violence against women, all around the world. It also has significant repercussions for women's health, yet, in some parts of the world, considered an acceptable practice within intimate partner relationships. Community-based interventions, on the other hand, offer promises as a strategy that can get community members involved in working to prevent IPV. This study evaluated a community mobilisation intervention to challenge attitudes toward IPV and prevent violence within intimate relationships.

Methods:

This mixed-method randomised community trial was conducted in selected rural communities in Oyo State, Nigeria, between January 2018 and April 2021. It employed a six-month community mobilisation intervention focused on creating awareness and challenging harmful social norms relating to IPV. In-depth interviews, focus group discussions and two cross-sectional surveys were conducted among men and women of reproductive age who were married at baseline and end line to estimate changes in key outcomes. Difference-in-difference regression models were estimated to compare changes in IPV levels in the intervention and control arms.

Conclusion:

This trial should demonstrate the effectiveness of community mobilisation interventions to change attitudes supportive of IPV and prevent women's experience of IPV.

DETAILED DESCRIPTION:
Background: Intimate partner violence (IPV) is arguably the most pernicious, pervasive, and persistent form of violence against women worldwide. It is an abuse of women's fundamental human rights and a public health concern. Experience of IPV by women has been associated with a mixture of both noticeable and frequently unnoticed outcomes, negatively affecting their health and wellbeing.

The prevalence of IPV is high in sub-Saharan Africa, where it is considered an element of the unwritten rules underpinning intimate relationships. Interventions that challenge these social norms are still evolving; community mobilization interventions, on the other hand, offer some potential in moderating the attitudes that permit or promote IPV. This study evaluated the effect of a community mobilization intervention on attitudes toward social norms that influence IPV in selected rural communities of Oyo State, Nigeria.

Methods: In a randomised community trial conducted in 8 rural communities of Oyo State, Nigeria, a six-month community mobilization intervention that consisted of advocacy to stakeholders, community workshops and small group discussions in 6 selected communities was tested compared with no intervention in the 2 control communities.

To engender community participation and sustainability of the intervention the investigator recruited and trained members of the community as 'Model Couples'. Community leaders, community health workers were also engaged to speak against IPV. Both the 'Model couples' and community leaders addressed topics like gender and power dynamics, IPV and its consequences, law prohibiting all forms of violence against women, social norms that influence IPV, and need to take action for change.

The intervention was tested among women of reproductive age, using a convergent parallel mixed-methods design. The study outcomes were attitudes toward social norms associated with IPV and experience of IPV. For the collection of quantitative data, a modified WHO women's health questionnaire was used, while an interview guide was developed for the collection of the qualitative data.

Conclusion: This trial should show community mobilization intervention as a strategy that can reduce women's experience of IPV and change attitudes toward IPV.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 59 years
* Women aged 18 to 49 years
* Currently married or cohabiting with a partner
* had lived in the community for a minimum of one year.

Exclusion Criteria:

* Married/ cohabiting males or females
* does not speak either Yoruba or English

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2650 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Attitudes towards social norms around intimate partner violence | One year before the survey
  Respondent agreed that a man is justified to beat his wife in seven scenarios provided. A score of 0 showed not supportive of physical IPV, while a score of 1 -7 showed attitude supportive of IPV

SECONDARY OUTCOMES:
Experience of intimate partner violence | One year before the survey
  Respondent answered yes to being physically, emotionally or sexually abused. A score of 0 showed no experience of IPV but a sore of more than 0 showed experience of IPV
Perpetration of intimate partner violence | One year before the survey
  Respondent answered yes to physically, emotionally or sexually abusing his wife. A score of 0 showed no perpetration of IPV but a sore of more than 0 showed perpetration of IPV
Community response to women's experience of of intimate partner violence | One year
  Community member agreed to intervening when they witnessed violence between couple

CONTACTS AND LOCATIONS:
Locations (1):
- Oriire LGA, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No